CLINICAL TRIAL: NCT03004729
Title: Symptoms Based Awareness Confirmation Study - CoMiSS Validation
Acronym: MOSAIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 16.05.CLI
Record Dates: First submitted 2016-11-24; First posted 2016-12-29 (Estimated); Last update posted 2018-08-20 (Actual); Status verified 2018-08

CONDITIONS: Cow Milk Allergy
Keywords: Allergy; Atopic Dermatitis; Immunoglobulin E (IgE); CMPA
MeSH Terms: conditions — Milk Hypersensitivity; Hypersensitivity; Dermatitis, Atopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CoMiSS (Other): Measure of CoMiSS followed by two weeks eviction Cow's milk protein diet and second CoMiSS measurement.
  Interventions: Other: CoMiSS questionnaire

INTERVENTIONS:
Other: CoMiSS questionnaire

SUMMARY:
The Cow's Milk-related Symptom Score (CoMiSS) tool has been developed to define a score to recognize cow's milk related symptoms in infants and young children.

Many infants and toddlers with symptoms that can be related to intake of cow's milk and cow's milk protein allergy (CMPA) are often not diagnosed due to the lack of specific markers.

The goal of this trial is to validate the CoMiSS tool in infants suspected of CMPA and investigate if the CoMiSS tool could be an alternative to the open challenge test needed to confirm the diagnosis of Cow Milk Protein Allergy.

ELIGIBILITY:
Inclusion Criteria:

* Male or female infant aged up to 6 months old
* Has been fed exclusively on cow's milk infant formula for at least one week
* Has CMPA symptoms that have been present for at least one week, and that developed within the first two months of starting cow's milk infant formula
* In the opinion of the investigator, requires a two week elimination diet with Amino Acid Formula (AAF).
* Had a gestational age at birth of 37 to 42 weeks
* Had a birthweight of 2500 g to 4500 g
* Informed consent signed by both parents, liable parent or legal guardian (if applicable).

Exclusion Criteria:

* Has ever received either an extensively hydrolysed infant formula or an AAF prior to enrolment
* Has a fever above 38.5°C at enrolment
* Has ever experienced a medically diagnosed serious anaphylactic reaction
* Use of antibiotic drugs at enrolment. Infants may be enrolled if antibiotics have been stopped at least 7 days prior to enrolment. (Antibiotic treatment can be initiated during the study if an infant develops a condition after enrolment that requires antibiotic treatment).
* Infant with a health condition or family situation that makes the infant unsuitable to participate in the trial according to the opinion of the investigator
* Infant or infant's carers are unable to comply with trial procedures
* Currently participating or has participated in another clinical trial within 4 weeks prior to trial start.

Ages: 1 Day to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 300 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
The accuracy in terms of the Area Under Curve (AUC) of the Receiver Operating Characteristic (ROC) curve of the change in CoMiSS. | baseline, Week 2

SECONDARY OUTCOMES:
CoMiSS and component scores | baseline, Week 2, Week 4
Family history of atopy | baseline
Method of delivery at birth | baseline
Anthropometric measurements | baseline
Volume intake of Alfamino formula every day | baseline, week 2
Physician's assessment of the likelihood that a subject has CMPA | baseline, week 2
The result of Oral food Challenge (OFC) | week 2, Week 4
Compliance to elimination diet | week 2

CONTACTS AND LOCATIONS:
Overall Officials: Zhengyan Zhao, Prof, Principal Investigator — The Children's Hospital Zhejiang University School of Medicine (ZUCH)
Locations (10):
- China (10):
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Children's Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Children's Hospital of Fuzhou in Fujian province, Fuzhou, Fujian
  - The Second Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Children's hospital of Zhengzhou, Zhengzhou, Henan
  - Hunan Children's Hospital, Hunan, Hunan
  - Children's Hospital of Shanghai, Shanghai, Shanghai Municipality
  - Children's hospital of Shanxi Women health center of Shanxi, Taiyuan, Shanxi
  - The Children's Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Maternal and child health care hospital of guangdong province, Guangzhou

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Host A. Cow's milk protein allergy and intolerance in infancy. Some clinical, epidemiological and immunological aspects. Pediatr Allergy Immunol. 1994;5(5 Suppl):1-36. PMID 7704117
- [Background] Sampson HA. Food allergy. Part 1: immunopathogenesis and clinical disorders. J Allergy Clin Immunol. 1999 May;103(5 Pt 1):717-28. doi: 10.1016/s0091-6749(99)70411-2. PMID 10329801
- [Background] Bock SA. Prospective appraisal of complaints of adverse reactions to foods in children during the first 3 years of life. Pediatrics. 1987 May;79(5):683-8. PMID 3575022
- [Background] Host A, Halken S. A prospective study of cow milk allergy in Danish infants during the first 3 years of life. Clinical course in relation to clinical and immunological type of hypersensitivity reaction. Allergy. 1990 Nov;45(8):587-96. doi: 10.1111/j.1398-9995.1990.tb00944.x. PMID 2288394
- [Background] Schrander JJ, van den Bogart JP, Forget PP, Schrander-Stumpel CT, Kuijten RH, Kester AD. Cow's milk protein intolerance in infants under 1 year of age: a prospective epidemiological study. Eur J Pediatr. 1993 Aug;152(8):640-4. doi: 10.1007/BF01955238. PMID 8404966
- [Background] Vandenplas Y; Althera Study Group; Steenhout P, Grathwohl D. A pilot study on the application of a symptom-based score for the diagnosis of cow's milk protein allergy. SAGE Open Med. 2014 Feb 13;2:2050312114523423. doi: 10.1177/2050312114523423. eCollection 2014. PMID 26770708
- [Background] Vandenplas Y, Steenhout P, Planoudis Y, Grathwohl D; Althera Study Group. Treating cow's milk protein allergy: a double-blind randomized trial comparing two extensively hydrolysed formulas with probiotics. Acta Paediatr. 2013 Oct;102(10):990-8. doi: 10.1111/apa.12349. Epub 2013 Aug 5. PMID 23837862
- [Background] Vandenplas Y, Dupont C, Eigenmann P, Host A, Kuitunen M, Ribes-Koninckx C, Shah N, Shamir R, Staiano A, Szajewska H, Von Berg A. A workshop report on the development of the Cow's Milk-related Symptom Score awareness tool for young children. Acta Paediatr. 2015 Apr;104(4):334-9. doi: 10.1111/apa.12902. Epub 2015 Jan 29. PMID 25557474
- [Derived] Vandenplas Y, Zhao ZY, Mukherjee R, Dupont C, Eigenmann P, Kuitunen M, Ribes Koninckx C, Szajewska H, von Berg A, Bajerova K, Meyer R, Salvatore S, Shamir R, Jarvi A, Heine RG; MOSAIC Study Investigator Group. Assessment of the Cow's Milk-related Symptom Score (CoMiSS) as a diagnostic tool for cow's milk protein allergy: a prospective, multicentre study in China (MOSAIC study). BMJ Open. 2022 Feb 17;12(2):e056641. doi: 10.1136/bmjopen-2021-056641. PMID 35177461
- [Derived] Vandenplas Y, Mukherjee R, Dupont C, Eigenmann P, Host A, Kuitunen M, Ribes-Koninkx C, Shah N, Szajewska H, von Berg A, Heine RG, Zhao ZY; on behalf the Chinese CoMiSS Investigator Team.. Protocol for the validation of sensitivity and specificity of the Cow's Milk-related Symptom Score (CoMiSS) against open food challenge in a single-blinded, prospective, multicentre trial in infants. BMJ Open. 2018 May 17;8(5):e019968. doi: 10.1136/bmjopen-2017-019968. PMID 29773698